CLINICAL TRIAL: NCT04633707
Title: Adjunctive Bright Light Therapy for Patients With Depression at Different Time Period: A Randomized Double-Blind, Placebo-Controlled Trial
Brief Title: Adjunctive Bright Light Therapy for Patients With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Kangguang Lin, Director, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Guangzhou Brain Hospital BLT
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Depressive Disorder; Light Therapy
Keywords: Depression; Bright Light Therapy; Time Period
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adjunctive morning BLT group (Experimental): treat participants with adjunctive BLT in the morning
  Interventions: Device: adjunctive bright white light therapy in the morning
- Adjunctive afternoon BLT group (Experimental): treat participants with adjunctive BLT in the afternoon
  Interventions: Device: adjunctive bright white light therapy in the afternoon
- Adjunctive placebo therapy group (Placebo Comparator): treat participants with adjunctive dim red light in the afternoon
  Interventions: Device: adjunctive dim red light therapy in the afternoon

INTERVENTIONS:
Device: adjunctive bright white light therapy in the morning — the participants would receive adjunctive bright white light therapy in the morning (light intensity: 10000lux, color: white light, duration of each intervention session: 30min, time period: 7:00~9:00) for 6 weeks.
  Arms: Adjunctive morning BLT group
Device: adjunctive bright white light therapy in the afternoon — the participants would receive adjunctive bright white light therapy in the afternoon (light intensity: 10000lux, color: white light, duration of each intervention session: 30min, time period: 12:00~14:00) for 6 weeks.
  Arms: Adjunctive afternoon BLT group
Device: adjunctive dim red light therapy in the afternoon — the participants received dim red light therapy (light intensity: <100lux, color: dark red, duration of each intervention session: 30min, time period: 12:00~14:00) for 6 weeks.
  Arms: Adjunctive placebo therapy group

SUMMARY:
The study would enroll depressed adolescents and adults with bipolar I or II disorder or major depressive disorder who are receiving stable psychiatric medication (excluding patients with hypomania or mania, mixed symptoms, or rapid cycling). Participants would be randomly assigned to treatment with either 1,0000-lux bright white light therapy in the morning or 1,0000-lux bright white light therapy in the afternoon, or <100-lux dim red placebo light therapy in the afternoon (N=59 for each group). Participants would be treated for 6 weeks. Symptoms would be assessed every two weeks with the 24-items Hamilton Depression Scale, the Young Mania Rating Scale, and the Pittsburgh Sleep Quality Index; salivary melatonin and cortisol concentrations will be also measured.

DETAILED DESCRIPTION:
The investigators would divide the participants enrolled into three groups: adjunctive morning bright light therapy (BLT) group (light intensity: 10000lux, color: white light, duration of each intervention session: 30min, time period of intervention: 7:00~9:00 a.m.), adjunctive afternoon BLT group (light intensity: 10000lux, color: white light, duration of each intervention session: 30min, time period of intervention: 12:00~14:00 p.m.), adjunctive placebo therapy group (light intensity: <100lux, color: dark red, duration of each intervention session: 30min, time period of intervention: 12:00~14:00 p.m.).

ELIGIBILITY:
Inclusion Criteria:

* 12-75 years old
* Diagnosed using DSM-5 criteria based on the Structured Clinical Interview for Patient Edition (SCID-P) for adults or Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime version (Kiddie-SADS-PL) for adolescents for the diagnosis of bipolar I or II disorder or major depressive disorder
* 24-items Hamilton Depression Rating Scale score ≥ 20, Young Mania Rating Scale score < 6
* Participants with bipolar disorder taking at least one mood stabilizer, and the types of drugs have not changed in one week;
* Antidepressants can be taken, and the types of antidepressants have not changed in one week
* Low-dose benzodiazepines can be used, with a maximum of 2 mg of lorazepam equivalent per day
* Right-handed
* Primary school education or above
* Sign informed consents after a full explanation of this study.

Exclusion Criteria:

* A history of brain organic disease or severe traumatic brain injury and severe physical disease;
* Drug, alcohol or other psychoactive substance abusers
* Severe suicide risk;
* Received modified electric convulsion therapy (MECT) in the past three months
* Comorbid with ophthalmic diseases (cataract, macular degeneration, glaucoma, retinitis pigmentosa, etc.) and diseases affecting the retina (retinopathy, diabetes, herpes, etc.)
* Taking photosensitive drugs (phenothiazines, antimalarials, propranolol, melatonin, hypericum, stimulants or NSAIDs)

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
response rate | up to week 6
  Participants with a decrease in 24-items Hamilton Depression Scale (HDRS) score of 50% or more from baseline. HDRS is used to measure the depressive severity；its measured time range is within the past week. In this study, version of 24-items is used. The patients are depressed when the total score are greater than 19 points, and there are no depression when the total scores are less than points.

SECONDARY OUTCOMES:
manic/hypomanic conversion rate | week 2; week 4; week 6
  The Young Mania Rating Scale (YMRS) is used to assess manic/hypomanic symptoms and their severity; its measured time range is within the past week. The higher the score, the more severe the symptom. If the total score is greater than or equal to 20, manic episode is considered; if the total score is less than 6, it means there is no manic/hypomanic symptoms.
side effect | week 2; week 4;week 6
  record the possible adverse reactions
sleep quality | week 2; week 4;week 6
  Pittsburgh Sleep Quality Index (PSQI) is used to evaluate sleep quality for last month. It's made of 7 items; every item is scored 1-4 point. Total score is obtained by adding up the points of 7 items. Total score range is 0~21 point. The sleep quality is worse when the total score is higher.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Kangguang, MD;PHD, Principal Investigator — Guangzhou Psychiatric Hospital
Locations (1):
- Guangzhou Brain Hospital (Guangzhou Huiai Hospital), Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No